CLINICAL TRIAL: NCT06583317
Title: Recurrent Pneumonia in Children At Assiut University Children's Hospital
Brief Title: Recurrent Pneumonia in Children
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dalia Abdelnaser Marouf Ahmed, 71515,Assiut, Assiut University
Other Study IDs: pnemonia
Record Dates: First submitted 2024-09-01; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Pneumonia; Lower Respiratory Tract Infection; Chest Infection
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aimed to analyses the clinical characteristics, risk factors and underlying causes as predictors of recurrent pneumonia in children attending AUCH

DETAILED DESCRIPTION:
Pneumonia is defined as inflammation of lung parenchyma due to various pathogenic organisms including bacteria, viruses, fungi and parasites. The key symptom to suspect childhood pneumonia is tachypnea. The World Health Organization (WHO) has defined tachypnea as respiratory rate >60 breaths/min in infants less than 2 months, >50 in infants 2 -12 months and >40 in children 1 to 5 years and >20 in children >5 years of age [1]. WHO has categorized pneumonia in children under-five years of age into two categories, pneumonia and severe pneumonia. Tachypnea with or without chest retraction is categorized as pneumonia while tachypnea with any danger signs (unable to feed or drink, hypothermia, unconsciousness, convulsion, signs of hypoxia including cyanosis, grunting, groaning, head nodding) as severe pneumonia [1].

Pneumonia is a common and described as the overlooked killer of children[2] as killing 1.1-1.4 million children every year. It accounts for 17%-19% of all deaths amongst children under 5 years of age; the majority of them are in developing countries [3,4] .In Egypt, children under 5 years approximate 13.4% of the total population[4] and pneumonia constitutes 19% of under-five mortality[5].

Recurrent pneumonia (RP) is defined as at least two episodes of pneumonia in one year or three episodes ever, with intercritical radiographic clearing of densities [6]. Incidence data indicate that RP occurs in 7.7%-9% of all children with CAP [7,8,9,10,11,12]. As a result, RP represents a frequent presenting manifestation in the general pediatric practice and is a very common reason for referral to pediatric chest physicians [7]. Factors linked to these infections could be recurrent aspirations, congenital structural anomalies of pulmonary and cardiovascular systems, defects in the clearance of airway secretions and immunodeficiency [13]

ELIGIBILITY:
Inclusion Criteria:

* • All children more than 1 month and less than 18 years of age

  * All cases presented by picture of recurrent pneumonia in the form of as at least two episodes of pneumonia in one year or three episodes ever, with radiographic clearing of densities in between.

Exclusion Criteria:

* • All children less than 1 month and more than 18 years

  * Evidence of malignancies
  * Evidence of congenital immune deficiency
  * Cases refusing to participate in research.
  * Cases missed for follow up.

Ages: 30 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children with recurrent pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
To delineate risk factors of recurrent chest infection. | Baseline
  Characteristics of studied children in AUCH as in feeding, nutritional status and growth parameters.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nair H, Simoes EA, Rudan I, Gessner BD, Azziz-Baumgartner E, Zhang JSF, Feikin DR, Mackenzie GA, Moiisi JC, Roca A, Baggett HC, Zaman SM, Singleton RJ, Lucero MG, Chandran A, Gentile A, Cohen C, Krishnan A, Bhutta ZA, Arguedas A, Clara AW, Andrade AL, Ope M, Ruvinsky RO, Hortal M, McCracken JP, Madhi SA, Bruce N, Qazi SA, Morris SS, El Arifeen S, Weber MW, Scott JAG, Brooks WA, Breiman RF, Campbell H; Severe Acute Lower Respiratory Infections Working Group. Global and regional burden of hospital admissions for severe acute lower respiratory infections in young children in 2010: a systematic analysis. Lancet. 2013 Apr 20;381(9875):1380-1390. doi: 10.1016/S0140-6736(12)61901-1. Epub 2013 Jan 29. PMID 23369797
- [Background] Bhutta ZA, Das JK, Walker N, Rizvi A, Campbell H, Rudan I, Black RE; Lancet Diarrhoea and Pneumonia Interventions Study Group. Interventions to address deaths from childhood pneumonia and diarrhoea equitably: what works and at what cost? Lancet. 2013 Apr 20;381(9875):1417-1429. doi: 10.1016/S0140-6736(13)60648-0. Epub 2013 Apr 12. PMID 23582723